CLINICAL TRIAL: NCT04609111
Title: ShorT and OPtimal Duration of Dual AntiPlatelet Therapy Study After Everolimus-eluting Cobalt-chromium Stent-3
Brief Title: ShorT and OPtimal Duration of Dual AntiPlatelet Therapy-3 Study
Acronym: STOPDAPT-3
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Study Statistician, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y0080
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome
Keywords: stent; percutaneous coronary transluminal angioplasty; bleeding; antiplatelet agents
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage | interventions — N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No aspirin (Active Comparator): To start prasugrel monotherapy before the index percutaneous coronary intervention (PCI) and to change into clopidogrel monotherapy at 1-month after the PCI.
  Interventions: Drug: No aspirin
- 1-month DAPT (Active Comparator): To start dual antiplatelet therapy comprising of aspirin and prasugrel before the index percutaneous coronary intervention (PCI) and to change into aspirin monotherapy at 1-month after the PCI.
  Interventions: Drug: 1-month DAPT

INTERVENTIONS:
Drug: No aspirin — 1-month prasugrel monotherapy followed by clopidogrel monotherapy
  Arms: No aspirin
Drug: 1-month DAPT — 1-month dual antiplatelet therapy comprising of aspirin and prasugrel followed by aspirin monotherapy
  Arms: 1-month DAPT

SUMMARY:
The purpose of this study is to explore the benefit of the prasugrel monotherapy without aspirin as compared with the 1-month dual therapy with aspirin and prasugrel in terms of reducing bleeding events after percutaneous coronary intervention (PCI) using cobalt-chromium everolimus-eluting stents (CoCr-EES, XienceTM) in patients with high bleeding risk or under the acute coronary syndrome patients.

DETAILED DESCRIPTION:
In the previous trial, 1-month dual antiplatelet therapy (DAPT) followed by clopidogrel monotherapy provided a net clinical benefit for the cardiovascular and bleeding events over 12-month DAPT with aspirin and clopidogrel after cobalt-chromium everolimus-eluting stent (CoCr-EES) implantation. However, even with very short DAPT, the rate of bleeding at 1-year remained very high in other trials that enrolled the patients with high bleeding risk (HBR). Notably, the risk of bleeding in patients with high bleeding risk (HBR) was particularly high within 1-month after percutaneous coronary intervention (PCI) in previous cohort data, when DAPT is implemented even in very short DAPT regimen. More recently, in another trial, prasugrel monotherapy without aspirin immediately after successful stent implantation was associated with no stent thrombosis in selected patients with low risk stable coronary artery disease. Aspirin-free strategy might be particularly beneficial in reducing bleeding in HBR patients. Patients with acute coronary syndrome (ACS) are also reported to be associated with higher risk for bleeding.

Therefore, we have planned a study to compare the cardiovascular and bleeding events at 1-month after PCI using CoCr-EES between no DAPT strategy and 1-month DAPT strategy in patients with HBR or ACS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to have percutaneous coronary intervention with exclusive use of everolimus-eluting stent (XienceTM series).
* Patients with high bleeding risk defined by Academic Research Consortium or acute coronary syndrome
* Patients who could take dual antiplatelet therapy with aspirin and P2Y12 inhibitors for 1-month

Exclusion Criteria:

* Patients who are judged to be unsuitable for participation by the principal investigator and co-investigator
* Patients with a known allergy to the study drugs
* Patients enrolled in the ongoing prospective interventional studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6002 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major bleeding | 1 month
  Bleeding defined as BARC criteria 3 or 5
Cardiovascular composite endpoint | 1 month
  Composite of cardiovascular death, myocardial infarction, ischemic stroke ,or definite stent thrombosis

SECONDARY OUTCOMES:
Death | 1 month
  Death from any cause
Death | 12 months
  Death from any cause
Cardiovascular death | 1 month
  Death from cardiac or vascular disease
Cardiovascular death | 12 months
  Death from cardiac or vascular disease
Myocardial infarction | 1 month
  Defined by arterial revascularization therapies study (ARTS) criteria
Myocardial infarction | 12 months
  Defined by arterial revascularization therapies study (ARTS) criteria
Stroke | 1 month
  Including both ischemic and hemorrhagic stroke
Stroke | 12 months
  Including both ischemic and hemorrhagic stroke
Ischemic stroke | 1 month
  Ischemic stroke with symptom lasting over 24 hours
Ischemic stroke | 12 months
  Ischemic stroke with symptom lasting over 24 hours
Hemorrhagic stroke | 1 month
  Intracerebral hemorrhage or subarachnoidal hemorrhage not associated with trauma
Hemorrhagic stroke | 12 months
  Intracerebral hemorrhage or subarachnoidal hemorrhage not associated with trauma
Stent thrombosis | 1 month
  Stent thrombosis defined by Academic Research Consortium definition
Stent thrombosis | 12 months
  Stent thrombosis defined by Academic Research Consortium definition
Target lesion failure | 1 month
  The angiographical confirmation of the restenosis of the target lesions
Target lesion failure | 12 months
  The angiographical confirmation of the restenosis of the target lesions
Target vessel failure | 1 month
  The angiographical confirmation of the restenosis or new lesion(s) of the target vessels or myocardial infarction involving the territory of target vessels
Target vessel failure | 12 months
  The angiographical confirmation of the restenosis or new lesion(s) of the target vessels or myocardial infarction involving the territory of target vessels
Any target lesion revascularization | 1 month
  Revascularization to the target lesions (including 5mm of both ends of the stent(s)) regardless percutaneous coronary intervention or coronary artery bypass grafting
Any target lesion revascularization | 12 months
  Revascularization to the target lesions (including 5mm of both ends of the stent(s)) regardless percutaneous coronary intervention or coronary artery bypass grafting
Clinically-driven target lesion revascularization | 1 month
  Target lesion revascularization with the anginal symptoms or the positive test for ischemia
Clinically-driven target lesion revascularization | 12 months
  Target lesion revascularization with the anginal symptoms or the positive test for ischemia
Non-target lesions revascularization | 1 month
  Revascularization to non-target lesions regardless percutaneous coronary intervention or coronary artery bypass grafting
Non-target lesions revascularization | 12 months
  Revascularization to non-target lesions regardless percutaneous coronary intervention or coronary artery bypass grafting
Coronary artery bypass grafting | 1 month
  Any coronary artery bypass grafting
Coronary artery bypass grafting | 12 months
  Any coronary artery bypass grafting
Any target vessel revascularization | 1 month
  Revascularization to the target vessel
Any target vessel revascularization | 12 months
  Revascularization to the target vessel
Any coronary revascularization | 1 month
  Revascularization regardless of percutaneous coronary intervention or coronary artery bypass grafting
Any coronary revascularization | 12 months
  Revascularization regardless of percutaneous coronary intervention or coronary artery bypass grafting
Type 2 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 1 month
  Type 2 bleeding defined by BARC criteria
Type 2 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 2 bleeding defined by BARC criteria
Type 3 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 1 month
  Type 3 bleeding defined by BARC criteria
Type 3 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 3 bleeding defined by BARC criteria
Type 4 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 1 month
  Type 4 bleeding defined by BARC criteria
Type 4 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 4 bleeding defined by BARC criteria
Type 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 1 month
  Type 5 bleeding defined by BARC criteria
Type 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 5 bleeding defined by BARC criteria
Type 2, 3, or 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 1 month
  Type 2, 3, or 5 bleeding defined by BARC criteria
Type 2, 3, or 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 2, 3, or 5 bleeding defined by BARC criteria
Major bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 1 month
  Major bleeding defined by TIMI criteria
Major bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 12 months
  Major bleeding defined by TIMI criteria
Minor bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 1 month
  Minor bleeding defined by TIMI criteria
Minor bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 12 months
  Minor bleeding defined by TIMI criteria
Major or minor bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 1 month
  Major or minor defined by TIMI criteria
Major or minor bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 12 months
  Major or minor defined by TIMI criteria
Severe bleeding in Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria | 1 month
  Severe bleeding defined by GUSTO criteria
Severe bleeding in Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria | 12 months
  Severe bleeding defined by GUSTO criteria
Moderate bleeding in Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria | 1 month
  Moderate bleeding defined by GUSTO criteria
Moderate bleeding in Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria | 12 months
  Moderate bleeding defined by GUSTO criteria
Moderate or severe bleeding in Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria | 1 month
  Moderate or severe bleeding defined by GUSTO criteria
Moderate or severe bleeding in Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria | 12 months
  Moderate or severe bleeding defined by GUSTO criteria
Intracranial bleeding | 1 month
  Intracranial bleeding regardless of spontaneous or trauma
Intracranial bleeding | 12 months
  Intracranial bleeding regardless of spontaneous or trauma
Gastrointestinal bleeding | 1 month
  Bleeding from gastrointestinal tract regardless of severity
Gastrointestinal bleeding | 12 months
  Bleeding from gastrointestinal tract regardless of severity
Gastrointestinal complaints | 1 month
  Requirement of upper gastric fiberscopy to examine the gastrointestinal complaints
Gastrointestinal complaints | 12 months
  Requirement of upper gastric fiberscopy to examine the gastrointestinal complaints

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nishikura T, Yamamoto K, Wakabayashi K, Natsuaki M, Watanabe H, Morimoto T, Obayashi Y, Nishikawa R, Kimura T, Ando K, Suwa S, Isawa T, Takenaka H, Ishikawa T, Onishi Y, Hibi K, Kawai K, Murakami T, Takasaki A, Higashitani N, Nakano M, Ono K, Kimura T; STOPDAPT-3 investigators. Effect of Proton Pump Inhibitors in Patients Undergoing Percutaneous Coronary Intervention With Aspirin-Free Strategy. JACC Asia. 2025 Nov 13:S2772-3747(25)00542-3. doi: 10.1016/j.jacasi.2025.09.015. Online ahead of print. PMID 41307518
- [Derived] Natsuaki M, Watanabe H, Morimoto T, Yamamoto K, Obayashi Y, Nishikawa R, Kimura T, Ando K, Suwa S, Isawa T, Takenaka H, Ishikawa T, Tamura T, Kawahatsu K, Hayashi F, Akao M, Serikawa T, Mori H, Kawamura T, Hagikura A, Shibata N, Ono K, Kimura T. Aspirin Versus Clopidogrel Beyond 1 Month After PCI in Patients With Oral Anticoagulation. Circ Cardiovasc Interv. 2025 Nov;18(11):e015495. doi: 10.1161/CIRCINTERVENTIONS.125.015495. Epub 2025 Sep 24. PMID 40988628
- [Derived] Obayashi Y, Natsuaki M, Watanabe H, Morimoto T, Yamamoto K, Nishikawa R, Kimura T, Ando K, Suwa S, Isawa T, Takenaka H, Ishikawa T, Tokuyama H, Sakamoto H, Fujita T, Nanasato M, Okayama H, Nishikura T, Kirigaya H, Nishida K, Ono K, Kimura T; STOPDAPT-3 Investigators. Aspirin vs Clopidogrel 1 Month After Acute Coronary Syndrome With High-Bleeding Risk or ST-Segment Elevation. JACC Cardiovasc Interv. 2025 Sep 8;18(17):2120-2135. doi: 10.1016/j.jcin.2025.03.029. Epub 2025 Jun 4. PMID 40471776
- [Derived] Ishikawa T, Natsuaki M, Watanabe H, Morimoto T, Yamamoto K, Obayashi Y, Nishikawa R, Ando K, Suwa S, Isawa T, Takenaka H, Yoshida R, Suzuki H, Nakazawa G, Kusuyama T, Morishima I, Hojo S, Tsutsumi J, Yamamoto H, Ueda H, Ono K, Kimura T. Aspirin-Free Strategy for PCI in Patients With High Bleeding Risk With or Without Acute Coronary Syndrome: A Subgroup Analysis From the STOPDAPT-3 Trial. Circ Cardiovasc Interv. 2025 Jul;18(7):e015197. doi: 10.1161/CIRCINTERVENTIONS.124.015197. Epub 2025 May 14. PMID 40365675
- [Derived] Domei T, Yamamoto K, Natsuaki M, Watanabe H, Morimoto T, Obayashi Y, Nishikawa R, Kimura T, Ando K, Suwa S, Isawa T, Takenaka H, Ishikawa T, Tamura T, Kawahatsu K, Hayashi F, Abe M, Serikawa T, Mori H, Kawamura T, Hagikura A, Shibata N, Ono K, Kimura T. Aspirin vs. clopidogrel monotherapy beyond 1 month after complex percutaneous coronary intervention: a pre-specified subgroup analysis of the STOPDAPT-3 trial. Eur Heart J Cardiovasc Pharmacother. 2025 Mar 13;11(2):198-209. doi: 10.1093/ehjcvp/pvaf002. PMID 39863419
- [Derived] Watanabe H, Natsuaki M, Morimoto T, Yamamoto K, Obayashi Y, Nishikawa R, Kimura T, Ando K, Domei T, Suwa S, Ogita M, Isawa T, Takenaka H, Yamamoto T, Ishikawa T, Hisauchi I, Wakabayashi K, Onishi Y, Hibi K, Kawai K, Yoshida R, Suzuki H, Nakazawa G, Kusuyama T, Morishima I, Ono K, Kimura T. Aspirin vs. clopidogrel monotherapy after percutaneous coronary intervention: 1-year follow-up of the STOPDAPT-3 trial. Eur Heart J. 2024 Dec 16;45(47):5042-5054. doi: 10.1093/eurheartj/ehae617. PMID 39215959
- [Derived] Watanabe H, Natsuaki M, Morimoto T, Yamamoto K, Obayashi Y, Nishikawa R, Hamatani Y, Ando K, Domei T, Suwa S, Ogita M, Isawa T, Takenaka H, Yamamoto T, Ishikawa T, Hisauchi I, Wakabayashi K, Onishi Y, Hibi K, Kawai K, Yoshida R, Suzuki H, Nakazawa G, Kusuyama T, Morishima I, Ono K, Kimura T; STOPDAPT-3 Investigators. Post-procedural Anticoagulation With Unfractionated Heparin in Acute Coronary Syndrome: Insight from the STOPDAPT-3 Trial. Am J Cardiol. 2024 Sep 1;226:83-96. doi: 10.1016/j.amjcard.2024.07.002. Epub 2024 Jul 6. PMID 38972535
- [Derived] Yamamoto K, Natsuaki M, Watanabe H, Morimoto T, Obayashi Y, Nishikawa R, Ando K, Suwa S, Isawa T, Takenaka H, Ishikawa T, Tamura T, Kawahatsu K, Hayashi F, Akao M, Serikawa T, Mori H, Kawamura T, Hagikura A, Shibata N, Ono K, Kimura T; STOPDAPT-3 Investigators. An Aspirin-Free Strategy for Immediate Treatment Following Complex Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2024 May 13;17(9):1119-1130. doi: 10.1016/j.jcin.2024.03.017. PMID 38749592
- [Derived] Natsuaki M, Watanabe H, Morimoto T, Yamamoto K, Obayashi Y, Nishikawa R, Ando K, Domei T, Suwa S, Ogita M, Isawa T, Takenaka H, Yamamoto T, Ishikawa T, Hisauchi I, Wakabayashi K, Onishi Y, Hibi K, Kawai K, Yoshida R, Suzuki H, Nakazawa G, Kusuyama T, Morishima I, Ono K, Kimura T. An Aspirin-Free Versus Dual Antiplatelet Strategy for Coronary Stenting: STOPDAPT-3 Randomized Trial. Circulation. 2024 Feb 20;149(8):585-600. doi: 10.1161/CIRCULATIONAHA.123.066720. Epub 2023 Nov 23. PMID 37994553